CLINICAL TRIAL: NCT07305909
Title: Two- and Three-Dimensional Quantification of Facial Symmetry Following Fat Grafting Versus Free Flap Reconstruction in Hemifacial Atrophy: A Retrospective Observational Study
Brief Title: Two- and Three-Dimensional Quantification of Facial Symmetry After Fat Grafting and Free Flap Reconstruction in Hemifacial Atrophy
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College (Other)
Collaborators: The Plastic Surgery Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Xiaolei Jin, Chief Physician, Professor of Plastic Surgery, Peking Union Medical College
Other Study IDs: 2024-344; 2024-344 (Other: Institutional Review Board of the Plastic Surgery Hospital, Chinese Academy of Medical Sciences)
Record Dates: First submitted 2025-12-13; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Hemifacial Atrophy
MeSH Terms: conditions — Facial Hemiatrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fat Grafting: Patients with hemifacial atrophy who underwent autologous fat grafting as the initial soft-tissue augmentation procedure. Outcomes were assessed preoperatively and at the first follow-up visit occurring ≥6 months postoperatively.
- Free Flap Reconstruction (ALT): Patients with hemifacial atrophy who underwent anterolateral thigh (ALT) free-flap reconstruction as the initial soft-tissue augmentation procedure. Outcomes were assessed preoperatively and at the first follow-up visit occurring ≥6 months postoperatively.

SUMMARY:
Hemifacial atrophy causes one side of the face to become smaller, leading to facial asymmetry. Surgeons often restore facial volume using either autologous fat grafting or free-flap reconstruction. However, it is not fully clear how much facial symmetry improves after surgery when measured objectively using two-dimensional (2D) photographs and three-dimensional (3D) surface scans.

This is a single-center, retrospective observational study of patients with hemifacial atrophy treated between January 2020 and December 2023 at [Plastic Surgery Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College]. We will quantify facial symmetry before surgery and at the first follow-up visit occurring at or beyond 6 months after the initial surgery. Symmetry outcomes will be assessed using standardized 2D photographs for all included patients, and 3D surface scans for a subset of patients. Complications will also be assessed at the first ≥6-month follow-up visit. We will compare changes in symmetry between patients treated with fat grafting and those treated with free-flap reconstruction.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of hemifacial atrophy (Parry-Romberg syndrome).

Underwent initial soft-tissue augmentation with either autologous fat grafting or free-flap reconstruction at the study center between January 2020 and December 2023.

Availability of standardized preoperative assessment and postoperative assessment at the first follow-up visit occurring ≥6 months after surgery (2D photographs required).

Exclusion Criteria:

Follow-up <6 months after the initial surgery.

Missing key imaging/photographic data required for outcome assessment.

Any additional facial augmentation or revision procedure performed before the first ≥6-month follow-up visit.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hemifacial atrophy treated at a single center between January 2020 and December 2023 who underwent initial facial volume restoration using autologous fat grafting or free-flap reconstruction. Outcomes were assessed preoperatively and at the first follow-up visit ≥6 months postoperatively. Three-dimensional surface scan analysis was performed in a subset with available 3D data.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Change in 2D Facial Symmetry Ratio | Baseline (preoperative) and first follow-up visit 6 months postoperatively
  Facial symmetry ratio calculated from standardized frontal 2D photographs using computerized photogrammetric analysis. The primary endpoint is the change from preoperative baseline to the first postoperative follow-up visit occurring at or beyond 6 months after the initial surgery.

SECONDARY OUTCOMES:
Change in 3D Volumetric Discrepancy Between Hemifaces | Baseline (preoperative) and first follow-up visit 6 months postoperatively
  Three-dimensional (3D) volumetric discrepancy between the affected and unaffected hemiface measured from 3D surface scans in the subset of participants with available 3D data. Change from baseline to the first ≥6-month follow-up visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Plastic Surgery Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality, China